CLINICAL TRIAL: NCT02283892
Title: Randomized Clinical Trial of the Impact of a Respiratory Complaints Assessment Checklist on Resources Utilization and Clinical Outcomes in an Acute Evaluation Outpatient Clinic
Brief Title: Respiratory Complaints Checklist Trial
Acronym: RCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, André Luis Ferreira Azeredo-Da-Silva, Internal Medicine Department Physician, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-0198
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Dyspnea; Cough
Keywords: respiratory complaints; dyspnea; cough; checklist
MeSH Terms: conditions — Dyspnea; Cough | interventions — Checklist; Clinical Protocols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Checklist (Experimental): 2 checklists available for consultation by the attending physician: (1) dyspnea evaluation checklist and (2) cough evaluation checklist. The checklists are available on computers and mobile devices (smartphone, PDA or tablet computer).
  Interventions: Other: Checklist
- Conventional assessment (Active Comparator): Evaluation of patients reporting dyspnea or cough made by the attending physician, without the use of the checklists for dyspnea or cough evaluation.
  Interventions: Other: Conventional evaluation

INTERVENTIONS:
Other: Checklist — 3 page checklist with suggestions of possible diagnosis according to clinical presentation of patients presenting with dyspnea or cough; also suggests diagnostic tests that are likely to be useful in each situation.
  Other Names: Clinical protocol
  Arms: Checklist
Other: Conventional evaluation — Physician evaluation without the use of checklists
  Other Names: Unaided physician evaluation
  Arms: Conventional assessment

SUMMARY:
This is a randomized clinical trial that evaluates the impact of using an internet-based checklist for systematic assessment of patients reporting respiratory complaints with the conventional assessment, without using the checklist.

DETAILED DESCRIPTION:
This is a randomized clinical trial that evaluates the impact of using an internet-based checklist for systematic assessment of patients reporting respiratory complaints with the conventional assessment, without using the checklist.

Study setting: emergency department related acute evaluation outpatient clinic

Inclusion criteria: 18 years of age or older; patients presenting to the ED reporting cough or dyspnea;

Exclusion criteria: acute respiratory failure; SpO2 < 92%; any signs of hemodynamic or respiratory instability; possible concurrent diagnosis requiring immediate assessment (e.g..: acute coronary syndrome or stroke; )

Primary outcome: need of reassessment in the ED or hospitalization within 1 month of index evaluation (intervention).

Secondary outcomes: number of complete blood counts ordered in the index evaluation; number of other diagnostic tests ordered in the index evaluation;

Randomization: block 1:1; stratified by gender and age (>50 years old).

Masking will be appllied to: patients; outcome assessors; data analysts;

ELIGIBILITY:
18 years of age or older; patients presenting to the ED reporting cough or dyspnea; legally capable.

Exclusion criteria: acute respiratory failure; SpO2 < 92%; any signs of hemodynamic or respiratory instability; possible concurrent diagnosis requiring immediate assessment (e.g..: acute coronary syndrome or stroke; )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Need to visit the emergency department or acute evaluation outpatient clinic | 1 month
Complete blood count ordered in the index evaluation | 1 month

SECONDARY OUTCOMES:
Number of diagnostic tests ordered in the index evaluation | 1 month
Hospital admission | 1 month
Antibiotics prescription | 1 month
  Frequency and type of antibiotic prescribed in each study arm
Major events | 1 month
  Composite endpoint: revisit to emergency department OR hospital admission OR death

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil